CLINICAL TRIAL: NCT04962568
Title: Ultrasonographic Evaluation of the Diaphragm During NHF Versus NIV Use in Respiratory Failure
Acronym: SENNI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jens Bräunlich (Other)
Responsible Party: Sponsor-Investigator, Jens Bräunlich, Sponsor and Investigator, Klinikum Emden
Organization: Klinikum Emden (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diaphragm Issues; Respiratory Failure With Hypoxia; Respiratory Failure With Hypercapnia; Non-invasive Mechanical Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHF-NIV (Experimental): Subjects will start with NHF. If all measurements are done, subjects will change to NIV. Same measurements will done.
  Interventions: Diagnostic Test: DTEE; Diagnostic Test: DTEI; Diagnostic Test: DEx
- NIV-NHF (Experimental): Subjects will start with NHF. If all measurements are done, subjects will change to NIV. Same measurements will done.
  Interventions: Diagnostic Test: DTEE; Diagnostic Test: DTEI; Diagnostic Test: DEx

INTERVENTIONS:
Diagnostic Test: DTEE — endexpiratory diaphragm thickness in mm
Diagnostic Test: DTEI — endinspiratory diaphragm thickness in mm
Diagnostic Test: DEx — diaphragm excursion during rest and diaphragmatic excursion during maximal inspiration in mm

SUMMARY:
This study will describe influence of NHF or NIV to different ultrasonographic parameters of the diaphragm. Therefor subjects will be randomized to the sequence NHF and than NIV or NIV and than NHF. In all subjects same parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* acute or chronic respiratory failure, hyperemic or hypercapnic
* age > 18 yrs
* written consent

Exclusion Criteria:

* critical disease (intubation, heart failure, lung edema,..)
* no compliance
* metabolic acidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2022-09-05 (Estimated)

PRIMARY OUTCOMES:
Changes in DTEE | 10 minutes
  Evaluation from baseline and between devices

SECONDARY OUTCOMES:
Changes in DTEI | 10 minutes
  Evaluation from baseline and between devices
Changes in Dex | 10 minutes
  Evaluation from baseline and between devices

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided